CLINICAL TRIAL: NCT02208362
Title: Phase I Study of Cellular ImmunoTx Using Memory Enriched T Cells Lentivirally Transduced to Express an IL13Rα2-Specific, Hinge-Optimized, 41BB-Costimulatory Chimeric Receptor and a Truncated CD19 for Pts With Rec/Ref MaligGlioma
Brief Title: Genetically Modified T-cells in Treating Patients With Recurrent or Refractory Malignant Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13384; NCI-2014-01488 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13384 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01FD005129 (FDA)
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Results first posted 2024-10-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Glioblastoma; Recurrent Malignant Glioma; Recurrent WHO Grade II Glioma; Recurrent WHO Grade III Glioma; Refractory Glioblastoma; Refractory Malignant Glioma; Refractory WHO Grade II Glioma; Refractory WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Tcm-derived CAR T cells, Intratumoral a/f biopsy [ICTb]) (Experimental): Arm 1 (Tcm-derived CAR T cells, Intratumoral a/f biopsy [ICTb]
  Interventions: Biological: Arm 1: IL13Ra2-specific CAR Tcm cells; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Quality-of-Life Assessment
- Arm 2 (Tcm-derived CAR T cells, ICTb/r) (Experimental): Arm 2 (Tcm-derived CAR T cells, Intratumoral a/f biopsy [ICTb] or Intracavitary a/f resection [ICTr])
  Interventions: Biological: Arm 2: IL13Ra2-specific CAR Tcm cells; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Quality-of-Life Assessment
- Arm 3 (Tcm-derived CAR T cells, Intraventricular [ICV]) (Experimental): Arm 3 (Tcm-derived CAR T cells, Intraventricular [ICV])
  Interventions: Biological: Arm 3: IL13Ra2-specific CAR Tcm cells; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Quality-of-Life Assessment
- Arm 4 (Tcm-derived CAR T cells, Dual delivery: both ICTb/r AND ICV) (Experimental): Arm 4 (Tcm-derived CAR T cells, Dual delivery: both ICTb/r AND ICV)
  Interventions: Biological: Arm 4: IL13Ra2-specific CAR Tcm cells; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Quality-of-Life Assessment
- Arm 5 (Tn/mem-derived CAR T cells, Dual delivery: both ICTb/r AND ICV) (Experimental): Arm 5 (Tn/mem-derived CAR T cells, Dual delivery: both ICTb/r AND ICV)
  Interventions: Biological: Arm 5: IL13Ra2-specific CAR Tn/mem cells; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Arm 1: IL13Ra2-specific CAR Tcm cells — Given via intratumoral catheter
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ Tcm-enriched T Cells; IL13Ra2-CAR/CD19t+ Tcm
  Arms: Arm 1 (Tcm-derived CAR T cells, Intratumoral a/f biopsy [ICTb])
Biological: Arm 2: IL13Ra2-specific CAR Tcm cells — Given via intratumoral/intracavitary catheter
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ Tcm-enriched T Cells; IL13Ra2-CAR/CD19t+ Tcm
  Arms: Arm 2 (Tcm-derived CAR T cells, ICTb/r)
Biological: Arm 3: IL13Ra2-specific CAR Tcm cells — Given via intraventricular catheter
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ Tcm-enriched T Cells; IL13Ra2-CAR/CD19t+ Tcm
  Arms: Arm 3 (Tcm-derived CAR T cells, Intraventricular [ICV])
Biological: Arm 4: IL13Ra2-specific CAR Tcm cells — Given via intratumoral or intracavitary, and via intraventricular catheter
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ Tcm-enriched T Cells; IL13Ra2-CAR/CD19t+ Tcm
  Arms: Arm 4 (Tcm-derived CAR T cells, Dual delivery: both ICTb/r AND ICV)
Biological: Arm 5: IL13Ra2-specific CAR Tn/mem cells — Given via intratumoral or intracavitary, and via intraventricular catheter
  Other Names: Autologous IL13(EQ)BBzeta/CD19t+ Tn/mem-enriched T Cells; IL13Ra2-CAR/CD19t+ Tn/mem
  Arms: Arm 5 (Tn/mem-derived CAR T cells, Dual delivery: both ICTb/r AND ICV)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Correlative studies
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; MRI Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging — Correlative studies
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of genetically modified T-cell immunotherapy in treating patients with malignant glioma that has come back (recurrent) or has not responded to therapy (refractory). A T cell is a type of immune cell that can recognize and kill abnormal cells in the body. T cells are taken from the patient's blood and a modified gene is placed into them in the laboratory and this may help them recognize and kill glioma cells. Genetically modified T-cells may also help the body build an immune response against the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility and safety of cellular immunotherapy utilizing ex vivo expanded autologous memory-enriched T cells (Arms 1, 2, 3, or 4 = Tcm or Arm 5 = Tn/mem) that are genetically modified using a self-inactivating (SIN) lentiviral vector to express an interleukin 13 receptor alpha 2 (IL13Ra2)-specific, hinge-optimized, 41BB-costimulatory chimeric antigen receptor (CAR), as well as a truncated CD19 (CD19t) for participants with recurrent/refractory malignant glioma in one of the following ways: (1) directly into the tumor (intratumoral), (2) into the tumor cavity (intracavitary), (3) into the lateral ventricles (intraventricular), or (4) into both the tumor/tumor cavity (intratumoral) and into the lateral ventricles (intraventricular) (dual delivery).

II. Determine maximum tolerated dose schedule (MTD)/maximum feasible dose schedule (MFD) and a recommended phase II dosing plan (RP2D) for each arm based on dose limiting toxicities (DLTs) and the full toxicity profile.

SECONDARY OBJECTIVES:

I. In research participants who receive the full schedule of three CAR+ T cell doses:

* Estimate disease response rates,
* Estimate median overall survival, and
* Estimate the mean change from baseline in quality of life using the EORTC QLQ-C30 during and post treatment;

II. Describe cytokine levels (tumor cavity fluid, CSF, peripheral blood) over the study period.

III. Describe CAR T cell and endogenous immune populations (CSF, tumor cavity fluid, peripheral blood) over the study period; and IV. Identify tumor and tumor micro-environment markers associated with response to CAR T cells.

EXPLORATORY OBJECTIVES:

I. Assess the timing and extent of brain inflammation following CAR T cell administration; II. Evaluate CAR T cell product characteristics; and

III. For research participants who undergo a second resection or autopsy:

* Evaluate CAR T cell persistence in the tumor micro-environment and the location of the CAR T cells with respect to the injection, and
* Evaluate IL13Rα2 antigen expression levels pre and post CAR T cell therapy.

OUTLINE: This is a dose-escalation study. Research subjects will receive an initial low dose (cycle 1) followed by 2 additional infusions at a higher cell dose (cycles 2 and 3) of autologous IL13Ra2-CAR/CD19t+ Tcm or Tn/mem, potentially followed by additional cycles at up to the highest tolerated cell dose (cycles 4+). CAR T cells will be administered in one of four ways:

ARM 1: (Intratumoral delivery a/f biopsy): Patients receive IL13Ra2-CAR/CD19t+ Tcm directly into the tumor via intratumoral (ICTb) catheter. Patients who progress on intratumoral administration may move to intraventricular catheter for the optional infusions.

ARM 2: (Intratumoral delivery a/f biopsy/Intracavitary a/f resection): Patients receive IL13Ra2-CAR/CD19t+ Tcm directly into the tumor via intratumoral (ICTb) catheter, or into the tumor resection cavity via intracavitary (ICTr) catheter. Patients who progress on intratumoral/intracavitary administration may move to intraventricular catheter for the optional infusions.

ARM 3: (Intraventricular delivery): Patients receive IL13Ra2-CAR/CD19t+ Tcm via intraventricular (ICV) catheter.

ARM 4: (Dual delivery): Patients receive IL13Ra2-CAR/CD19t+ Tcm via ICTb/r catheter and ICV catheter. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).

ARM 5: (Dual delivery): Patients receive IL13Ra2-CAR/CD19t+ Tn/mem via ICTb/r catheter and ICV catheter. Based on clinical response after the first 3 infusions, the study principal investigator may decide to continue with the optional infusions at either one or both sites (instead of requiring injections at both sites).

CAR T cells will be administered at one of three dose schedules:

* Dose Schedule 1: Cycle 1 - 2x106 CAR T cells, Cycle 2 & 3 - 10x106 CAR T cells, Total dose - 22x106 CAR T cells; Optional cycles ≤10x106 CAR T cells
* Dose Schedule 2: Cycle 1 - 10x106 CAR T cells, Cycle 2 & 3 - 50x106 CAR T cells, Total dose - 110x106 CAR T cells; Optional cycles ≤50x106 CAR T cells
* Dose Schedule 3: Cycle 1 - 20x106 CAR T cells, Cycle 2 & 3 - 100x106 CAR T cells, Total dose - 220x106 CAR T cells; Optional cycles ≤100x106 CAR T cells

After completion of the study treatment, patients are followed up at 4 weeks, 3, 6, 8, 10, and 12 months, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* SCREENING INCLUSION CRITERIA
* Participant has a prior histologically-confirmed diagnosis of a grade III or IV glioma, or has a prior histologically-confirmed diagnosis of a grade II glioma and now has radiographic progression consistent with a grade III or IV malignant glioma (MG) after completing standard therapy
* Radiographic evidence of progression/recurrence of the measurable disease more than 12 weeks after the end of the initial radiation therapy
* Karnofsky performance status (KPS) >= 60%
* Life expectancy > 4 weeks
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* City of Hope (COH) Clinical Pathology confirms IL13R alpha 2+ tumor expression by immunohistochemistry (>= 20%, 1+)
* All research participants must have the ability to understand and the willingness to sign a written informed consent
* ELIGIBILITY TO PROCEED WITH PERIPHERAL BLOOD MONONUCLEAR CELL (PBMC) COLLECTION
* Research participant must not require more than 2 mg three times daily (TID) of dexamethasone on the day of PBMC collection.
* Research participant must have appropriate venous access
* At least 2 weeks must have elapsed since the research participant received his/her last dose of prior chemotherapy or radiation
* ELIGIBILITY TO PROCEED WITH RICKHAM PLACEMENT
* Creatinine < 1.6 mg/dL
* White blood cell (WBC) > 2,000/dl or
* Absolute neutrophil count (ANC) > 1,000
* Platelets >= 100,000/dl
* International normalized ratio (INR) < 1.3
* Bilirubin < 1.5 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limits of normal
* An interval of at least 12 weeks must have elapsed since the completion of initial radiation therapy
* Wash-out requirements (standard or investigational):

  * At least 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen
  * At least 23 days since the completion of Temodar and/or 4 weeks for any other non-nitrosourea-containing cytotoxic chemotherapy regimen; if a patient's most recent treatment was with a targeted agent only, and s/he has recovered from any toxicity of this targeted agent, then a waiting period of only 2 weeks is needed from the last dose and the start of study treatment, with the exception of bevacizumab where a wash out period of at least 4 weeks is required before starting study treatment
* ELIGIBILITY FOR ENROLLMENT AND TO PROCEED WITH CAR T CELL INFUSION
* Research participant has a released cryopreserved T cell product
* Research participant does not require supplemental oxygen to keep saturation greater than 95% and/or does not have presence of any radiographic abnormalities on chest x-ray that are progressive
* Research participant does not require pressor support and/or does not have symptomatic cardiac arrhythmias
* Research participant does not have a fever exceeding 38.5° Celsius (C); there is an absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to T cell infusion and/or there aren't any indications of meningitis
* Research participant serum total bilirubin does not exceed 2 x normal limit
* Research participant transaminases does not exceed 2 x normal limit
* Research participant serum creatinine =< 1.8 mg/dL
* Research participant does not have uncontrolled seizure activity following surgery prior to starting the first T cell dose
* Research participant platelet count must be >= 100,000; however, if platelet level is between 75,000-99,000, then T-cell infusion may proceed after platelet transfusion is given and the post transfusion platelet count is >= 100,000
* Research participants must not require more than 2 mg TID of dexamethasone during T cell therapy

Exclusion Criteria:

* SCREENING EXCLUSION CRITERIA
* Research participant requires supplemental oxygen to keep saturation greater than 95% and the situation is not expected to resolve within 2 weeks
* Research participant requires pressor support and/or has symptomatic cardiac arrhythmias
* Research participant requires dialysis
* Research participant has uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study; a legal guardian may substitute for the research participant
* Research participants with any non-malignant intercurrent illness which is either poorly controlled with currently available treatment, or which is of such severity that the investigators deem it unwise to enter the research participant on protocol shall be ineligible
* Research participants with any other active malignancies
* Research participants being treated for severe infection or who are recovering from major surgery are ineligible until recovery is deemed complete by the investigator
* Research participants with any uncontrolled illness including ongoing or active infection; research participants with known active hepatitis B or C infection; research participants with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections
* Research participants who have confirmed human immunodeficiency virus (HIV) within 4 weeks of screening

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2026-06-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Badie, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Brown CE, Hibbard JC, Alizadeh D, Blanchard MS, Natri HM, Wang D, Ostberg JR, Aguilar B, Wagner JR, Paul JA, Starr R, Wong RA, Chen W, Shulkin N, Aftabizadeh M, Filippov A, Chaudhry A, Ressler JA, Kilpatrick J, Myers-McNamara P, Chen M, Wang LD, Rockne RC, Georges J, Portnow J, Barish ME, D'Apuzzo M, Banovich NE, Forman SJ, Badie B. Locoregional delivery of IL-13Ralpha2-targeting CAR-T cells in recurrent high-grade glioma: a phase 1 trial. Nat Med. 2024 Apr;30(4):1001-1012. doi: 10.1038/s41591-024-02875-1. Epub 2024 Mar 7. PMID 38454126
- [Derived] Brown CE, Alizadeh D, Starr R, Weng L, Wagner JR, Naranjo A, Ostberg JR, Blanchard MS, Kilpatrick J, Simpson J, Kurien A, Priceman SJ, Wang X, Harshbarger TL, D'Apuzzo M, Ressler JA, Jensen MC, Barish ME, Chen M, Portnow J, Forman SJ, Badie B. Regression of Glioblastoma after Chimeric Antigen Receptor T-Cell Therapy. N Engl J Med. 2016 Dec 29;375(26):2561-9. doi: 10.1056/NEJMoa1610497. PMID 28029927

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm 1 was biopsy only due to concern of potentially higher toxicity rates with increased tumor burden. After no dose-limiting toxicities were observed on Arm 1, dose schedule (DS)1, this Arm was closed and participants were included in the other dose schedules in Arm 2.
Groups:
- Arm 1 Dose Schedule 1: Intratumoral a/f biopsy [ICTb]
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral catheter weekly for 3 weeks
- Arm 2 Dose Schedule 1: CAR Tcm cells Intratumoral a/f biopsy [ICTb] or Intracavitary a/f resection [ICTr]
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter weekly for 3 weeks
- Arm 2 Dose Schedule 2: CAR Tcm cells Intratumoral a/f biopsy [ICTb] or Intracavitary a/f resection [ICTr]
  Dose schedule 2
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter weekly for 3 weeks
- Arm 2 Dose Schedule 3: CAR Tcm cells Intratumoral a/f biopsy [ICTb] or Intracavitary a/f resection [ICTr]
  Dose schedule 3
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter weekly for 3 weeks
- Arm 3 Dose Schedule 1: CAR Tcm cells intraventricular [ICV]
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intraventricular catheter weekly for 3 weeks
- Arm 3 Dose Schedule 2: CAR Tcm cells intraventricular [ICV]
  Dose schedule 2
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intraventricular catheter weekly for 3 weeks
- Arm 3 Dose Schedule 3: CAR Tcm cells intraventricular [ICV]
  Dose schedule 3
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intraventricular catheter weekly for 3 weeks
- Arm 4 Dose Schedule 1: CAR Tcm cells ICTb/r and ICV
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
- Arm 4 Dose Schedule 2: CAR Tcm cells ICTb/r and ICV
  Dose schedule 2
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
- Arm 5 Dose Schedule 1: CAR Tn/mem cells ICTb/r and ICV
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tn/mem cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
- Arm 5 Dose Schedule 2: CAR Tn/mem cells ICTb/r and ICV
  Dose schedule 2
  Patients receive IL13Ra2-CAR/CD19t+ Tn/mem cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
- Arm 5 Dose Schedule 3: CAR Tn/mem cells ICTb/r and ICV
  Dose schedule 3
  Patients receive IL13Ra2-CAR/CD19t+ Tn/mem cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
Period: Overall Study
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
Started | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 8 | 11
Completed | 2 | 3 | 4 | 10 | 3 | 3 | 4 | 3 | 5 | 3 | 7 | 11
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Not completed — Participant did not complete treatment | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Participant received disallowed treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 Dose Schedule 1: CAR Tcm cells Intratumoral a/f biopsy [ICTb]
  Dose schedule 1
  Patients receive IL13Ra2-CAR/CD19t+ Tcm cells via intratumoral or intracavitary catheter weekly for 3 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3 | Total
Number analyzed (Participants) | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 8 | 11 | 65
Age, Continuous [Median (Full Range); unit: years] | 52.5 [40 to 65] | 56 [38 to 67] | 55.5 [41 to 70] | 44 [32 to 71] | 56 [44 to 60] | 49 [42 to 57] | 56 [16 to 69] | 59.5 [54 to 65] | 53 [30 to 65] | 32 [32 to 35] | 49 [34 to 56] | 48 [25 to 65] | 49 [16 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 3 | 1 | 0 | 1 | 2 | 3 | 2 | 4 | 5 | 25
  Male | 1 | 1 | 4 | 7 | 2 | 3 | 4 | 2 | 5 | 1 | 4 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 11
  Not Hispanic or Latino | 1 | 3 | 4 | 8 | 3 | 3 | 5 | 4 | 7 | 3 | 4 | 6 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 4 | 3 | 10 | 3 | 3 | 5 | 3 | 6 | 2 | 6 | 8 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 8 | 11 | 65
Histology [Count of Participants; unit: Participants]
  Grade 4 glioblastoma IDH wildtype | 2 | 3 | 3 | 6 | 3 | 2 | 2 | 4 | 6 | 1 | 5 | 10 | 47
  Grade 4 diffuse midline glioma, H3 K27-altered | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Grade 3 astrocytoma, IDH mutant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Grade 3 oligodendroglioma, IDH-mutant and 1p/19q-codeleted | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
  Grade 3 supratentorial ependymoma, NEC | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Grade 4 diffuse astrocytoma, NOS | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Grade 4 astrocytoma, IDH mutant | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Toxicity Related to CAR T Cells
Description: Grade 3 or higher toxicity profile for adverse events probably or definitely related to CAR T cells as assessed by the NCI CTCAE version 4.0.
Time Frame: An average of 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
Number analyzed (Participants) | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 8 | 11
Participants
  Encephalopathy: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Encephalopathy: No | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 3 | 8 | 3 | 8 | 11
  Ataxia: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Ataxia: No | 2 | 4 | 4 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 8 | 10

2. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity (DLT)
Description: Toxicities will be graded using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A DLT is defined as events attributable to T-cell infusion (probable or definite) with a few expected events that resolve within a specified time and occurring from the time of initial CAR T cell infusion through 1 week following the last infusion cycle (not including optional cycles) unless otherwise specified in this definition:
  1. Two grade 3 toxicities at the same dose with the exception of those grade 3 toxicities listed below.
  2. Any grade 3 Cytokine release syndrome (CRS) toxicity lasting more than 72 hours without intervention
  3. Any grade 3 or higher allergic reaction
  4. Any grade 3 or higher autoimmune reaction
  5. Any grade 4 toxicity
Time Frame: Up to 1 week following the last course, up to a total of 4 weeks (not including optional courses 4-6)
Population: 11 total participants were deemed not eligible for dose escalation due to the following: 7 did not receive the full 3 cycles of CAR T, 1 had too much time between surgery and CAR T, 2 received disallowed treatment, and 1 did not receive their full treatment schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
Number analyzed (Participants) | 2 | 3 | 3 | 9 | 3 | 3 | 4 | 3 | 5 | 3 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Active Response Determined by Response Assessment in Neuro-Oncology (RANO) Criteria
Description: Counts of active response and progression determined by RANO. Participants achieving stable disease (SD), partial remission (PR), or complete remission (CR) are counted as active.
  RANO:
  Complete Response (CR): Disappearance of all enhancing disease sustained for 4 weeks, stable or improved FLAIR/T2 lesions, no new lesions, off corticosteroids and neurologically stable or improved.
  Partial Response (PR): At least a 50% decrease of all measurable enhancing lesions sustained for 4 weeks, no progression of non-measurable disease, stable or improved FLAIR/T2 lesions, no new lesions, corticosteroids dose stable or reduced and neurologically stable or improved.
  Stable Disease (SD): Does not qualify for CR, PR or PD, stable FLAIR/T2 lesions, stable or reduced corticosteroids, clinically stable Progressive Disease (PD): At least a 25% increase in enhancing lesions despite stable or increasing steroid dose, increase in FLAIR/T2 lesions, any new lesions, clinical deteriorations.
Time Frame: Between 4 and 8 weeks post 1st CAR T infusion
Population: 7 total participants were deemed not eligible for response due to the following: 5 did not receive the full 3 cycles of CAR T, 1 received disallowed treatment, and 1 did not receive their full treatment schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
Number analyzed (Participants) | 2 | 3 | 4 | 10 | 3 | 3 | 4 | 3 | 5 | 3 | 7 | 11
Participants
  Active | 0 | 2 | 3 | 5 | 1 | 2 | 2 | 1 | 2 | 0 | 3 | 8
  Progression | 2 | 1 | 1 | 5 | 2 | 1 | 2 | 2 | 3 | 3 | 4 | 3

4. Secondary Outcome: Number of Participants Alive at 6 Months
Description: Participants were assessed for vital status up to 6 months post surgery.
Time Frame: From surgery to death from any cause or six months, whichever occurred first
Population: 8 total participants were deemed not eligible for survival due to the following: 5 did not receive the full 3 cycles of CAR T, 1 received disallowed treatment, 1 had too much time between surgery and CAR T, and 1 did not receive their full treatment schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
Number analyzed (Participants) | 2 | 3 | 4 | 10 | 3 | 3 | 4 | 3 | 5 | 3 | 7 | 10
Participants | 1 | 2 | 2 | 6 | 2 | 3 | 3 | 1 | 2 | 2 | 5 | 8

ADVERSE EVENTS:
Time Frame: While on study, an average of 11 months
Groups:
- Arm 5 Dose Schedule 3: CAR Tn/mem cells ICTb/r and ICV
  Dose schedule3
  Patients receive IL13Ra2-CAR/CD19t+ Tn/mem cells via intratumoral or intracavitary catheter and intraventricular catheter weekly for 3 weeks
Arm/Group | Arm 1 Dose Schedule 1 | Arm 2 Dose Schedule 1 | Arm 2 Dose Schedule 2 | Arm 2 Dose Schedule 3 | Arm 3 Dose Schedule 1 | Arm 3 Dose Schedule 2 | Arm 3 Dose Schedule 3 | Arm 4 Dose Schedule 1 | Arm 4 Dose Schedule 2 | Arm 5 Dose Schedule 1 | Arm 5 Dose Schedule 2 | Arm 5 Dose Schedule 3
All-Cause Mortality (participants affected / at risk) | 2/2 | 4/4 | 4/4 | 10/10 | 3/3 | 2/3 | 4/5 | 4/4 | 7/8 | 3/3 | 5/8 | 11/11
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 2/4 | 2/10 | 3/3 | 0/3 | 3/5 | 3/4 | 4/8 | 2/3 | 5/8 | 5/11
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 4/4 | 10/10 | 3/3 | 3/3 | 5/5 | 4/4 | 8/8 | 3/3 | 8/8 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Dose Schedule 1 (N=2) | Arm 2 Dose Schedule 1 (N=4) | Arm 2 Dose Schedule 2 (N=4) | Arm 2 Dose Schedule 3 (N=10) | Arm 3 Dose Schedule 1 (N=3) | Arm 3 Dose Schedule 2 (N=3) | Arm 3 Dose Schedule 3 (N=5) | Arm 4 Dose Schedule 1 (N=4) | Arm 4 Dose Schedule 2 (N=8) | Arm 5 Dose Schedule 1 (N=3) | Arm 5 Dose Schedule 2 (N=8) | Arm 5 Dose Schedule 3 (N=11)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Encephalitis infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema cerebral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
tumor progression and cerebritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
L hemipheric subdural hydroma/hematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Dose Schedule 1 (N=2) | Arm 2 Dose Schedule 1 (N=4) | Arm 2 Dose Schedule 2 (N=4) | Arm 2 Dose Schedule 3 (N=10) | Arm 3 Dose Schedule 1 (N=3) | Arm 3 Dose Schedule 2 (N=3) | Arm 3 Dose Schedule 3 (N=5) | Arm 4 Dose Schedule 1 (N=4) | Arm 4 Dose Schedule 2 (N=8) | Arm 5 Dose Schedule 1 (N=3) | Arm 5 Dose Schedule 2 (N=8) | Arm 5 Dose Schedule 3 (N=11)
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 5 | 3 | 3 | 4 | 2 | 5 | 2 | 6 | 8
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 3 | 5 | 2 | 3 | 3 | 4 | 4 | 1 | 3 | 6
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 3 | 7 | 2 | 2 | 3 | 2 | 5 | 3 | 4 | 8
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
feeling of fullness in L ear (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
R ear feeling plugged after hyperbaric O2 tx. otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ear pressure (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ear congestion due to URI (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
"cloudiness" of vision, noted in OT only once (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
frequent blinking, a long term issue (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
visual disturbance (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
visual difficulty (not blurriness) (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
eye pressure (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
vision change (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
double vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
eyelid swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
vision impairment, L peripheral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
L visual peripheral field cut (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 2
mild chewing difficulty (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
canker sore (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cold Sore (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 3 | 4 | 3 | 5 | 8
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 2 | 4 | 3 | 2 | 7
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 2 | 7 | 0 | 3 | 3 | 2 | 3 | 2 | 4 | 8
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 4 | 9 | 3 | 3 | 4 | 4 | 8 | 3 | 7 | 10
Fever (General disorders) | 1 | 1 | 2 | 5 | 2 | 3 | 3 | 1 | 2 | 2 | 4 | 5
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 4 | 3
diaphoresis (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
profuse sweating only on L side (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
occ chest tightness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
night sweats (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
sweating (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
drowsiness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
diaphoresis during hypoglycemia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
bodyaches (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
cold intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
edema generalized (fluid retention) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 4
Pain (General disorders) | 2 | 0 | 0 | 2 | 3 | 2 | 0 | 1 | 2 | 2 | 3 | 1
Edema limbs (General disorders) | 1 | 1 | 2 | 5 | 2 | 2 | 3 | 2 | 2 | 0 | 1 | 1
Edema trunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
bacteremia, wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ventriculitis, wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peripheral nerve infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 4 | 2 | 1 | 2 | 0 | 2 | 2 | 3 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 1 | 3 | 1 | 3 | 5
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 4 | 1 | 3 | 3 | 0 | 2 | 3 | 4 | 2 | 5 | 3
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 3 | 3 | 1 | 1 | 2 | 1 | 4 | 1 | 3 | 2
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 2 | 2 | 2 | 1 | 0 | 2 | 2 | 4 | 2 | 4 | 3
Weight loss (Investigations) | 0 | 1 | 2 | 2 | 2 | 1 | 2 | 0 | 4 | 0 | 3 | 1
White blood cell decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 3 | 0 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 5 | 3 | 1 | 3 | 3 | 4 | 1 | 6 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 2 | 1 | 4 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 6 | 1 | 0 | 2 | 0 | 2 | 1 | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 5 | 1 | 2 | 1 | 2 | 4 | 2 | 6 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 5 | 3 | 0 | 4 | 3 | 6 | 2 | 7 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 2
Obesity (Metabolism and nutrition disorders) | 1 | 3 | 2 | 4 | 0 | 3 | 2 | 0 | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pain/clicking of R jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
compression fractures L spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
groin pain due to inguinal hernia; hernia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
inguinal hernia; hernia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
generalized body aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 0 | 2 | 2 | 1 | 1 | 3 | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 1 | 2 | 2 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 1 | 3 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 1 | 3 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
lump L temporal area (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 5
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 1 | 2 | 3 | 2 | 1 | 2 | 2 | 0 | 1 | 3 | 3
Edema cerebral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 7 | 3 | 3 | 5 | 4 | 7 | 3 | 8 | 9
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 3 | 4 | 3 | 2 | 2
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 0 | 2 | 3 | 1 | 7
Movements involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
tumor progression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
olfactory aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of coldness near right ear. Per patient, present since surgery (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
emotional instability (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
emotional lability (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
off balance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
other not specified (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
pseudomeningocele (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
L hand twitching, a long term issue (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
drooling when eating from L side of mouth (per pt) (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
L sided hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
decreased motor skills (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
slight balance issues (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
funny sensation on R side of mouth (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
subgaleal fluid collection (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 2
strange sensation/aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
steroid taper (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
L sided numbness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
shuffling steps/leaning forward (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
R hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
balance issues (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
altered mental status (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
illogical speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
facial twitching in AM (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
fog brain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
R leg paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
R ptosis after botox injection (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 3 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 3 | 2 | 1 | 4 | 3
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 5
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 2 | 3
Confusion (Psychiatric disorders) | 0 | 2 | 3 | 2 | 3 | 1 | 3 | 2 | 3 | 1 | 3 | 8
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 3 | 3 | 1 | 3 | 1 | 3 | 2 | 4 | 4
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
emotional lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 1
urinary/abdominal "pressure" due to UTI (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
urinary hesitancy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
difficulty urinating (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 2 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 5 | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
problems with mucous and sputum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pulmonary infiltrates, due to DVT/PE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
chest tightness, inhaler helped (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
rhinitis/coryza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
chest congestion. Poss due to pembro (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 1 | 1 | 2 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 1
skin erythema from suture abcess (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
wound drainage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
erythema over Rickham (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
groin skin tightness, due to steroids (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
redness at temporal Rickham (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
blistered skin under headwrap (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
skin tear on leg (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
swelling over Rickham (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
skin tear, R frontal scalp due to scrape (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
skin ulceration R foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
blister on finger due to burn from hot water (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
erythema - steroid use (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
redness at Rickham (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
itching at Rickham (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
erythema/redness on palms; cabozantanib (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 4 | 3 | 10 | 3 | 3 | 5 | 4 | 8 | 3 | 7 | 10
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT02208362/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02208362/ICF_001.pdf